CLINICAL TRIAL: NCT05681858
Title: Coronary Artery Plaque, Perivascular Inflammation and Myocardial Ischemia in Patients With Myocardial Infraction and Non-obstructive Coronary Arteries
Brief Title: Plaque Burden and Ischemia in MINOCA
Status: Recruiting | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Haraldsplass Deaconess Hospital (Other)
Responsible Party: Principal Investigator, Mai Tone Lønnebakken, Professor M.D., University of Bergen
Other Study IDs: 463549
Record Dates: First submitted 2023-01-03; First posted 2023-01-12 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: MINOCA
MeSH Terms: conditions — MINOCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT coronary angiography and [12N] NH3 PET-MR: All patients will undergo CT coronary angiography and stress [12N] NH3 PET-MR
  Interventions: Diagnostic Test: CT coronary angiography and [12N] NH3 PET-MR

INTERVENTIONS:
Diagnostic Test: CT coronary angiography and [12N] NH3 PET-MR — Advanced coronary artery plaque analysis, myocardial ischemia and coronary flow reserve

SUMMARY:
The goal of this clinical trial is to assess coronary artery plaque burden, perivascular inflammation and extent of myocardial ischemia in patients presenting with acute myocardial infarction and non-obstructive coronary artery disease. The main question it aims to answer are:

* Identify coronary artery anatomy, plaque burden, composition and high-risk plaque features by CT coronary angiography in MINOCA
* Assess presence, extent and severity of myocardial ischemia in MINOCA

Participants will examined by CT coronary angiography and stress [12N] NH3 PET-MR.

ELIGIBILITY:
Inclusion Criteria:

* Acute chest pain
* Elevated troponin
* Non-obstructive coronary arteries by coronary angiography

Exclusion Criteria:

* Obstructive coronary artery disease
* Contraindications against CT coronary angiography or stress [12N] NH3 PET-MR
* Not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with acute myocardial infarction and non-obstructive coronary artery disease by coronary angiography
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Plaque burden | 1 week
Myocardial ischemia | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Science, University of Bergen, Bergen, Norway